CLINICAL TRIAL: NCT01484990
Title: A Pharmacokinetic Study of Levodopa and Carbidopa Intestinal Gel in Subjects With Advanced Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S187.1.002; 2009-016837-84 (EudraCT Number)
Record Dates: First submitted 2011-07-28; First posted 2011-12-05 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2011-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; levodopa; carbidopa; Duodopa; intestinal gel
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Levodopa-Carbidopa

INTERVENTIONS:
Drug: Levodopa-Carbidopa — Intestinal Gel

SUMMARY:
A Pharmacokinetic Study of Levodopa and Carbidopa Intestinal Gel in Subjects with Advanced Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects at least 30 years old;
2. Subjects with advanced Parkinson's disease who are already on LCIG (Duodopa®) for at least 30 days;
3. Body mass index range from 18.0 to 30.0 kg/m2

Exclusion Criteria

1. Subjects who are considered to be violent or subjects considered at suicidal risk by the investigator;
2. Clinically significant abnormal laboratory data at baseline or any abnormal laboratory value that could interfere with the study assessments;
3. Subjects with serious symptomatic cerebral disease, cerebrovascular disease, focal neurological lesions (previous brain surgery), any acute brain trauma requiring treatment with anticonvulsant therapy, or acute stroke

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Profile of Pharmacokinetics | 5mins, then every 30 minutes up to 8 hours (0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8 hour), 12, 16 (immediately after flushing the tube), 17, 18, and 19 hours.
  Levodopa, Carbidopa and Metabolite:Cmax, Cmin, Area Under Curve, T max, half life, peak-trough fluctuation.
Safety and Tolerability Data Assessments (e.g., clinical laboratory tests, orthostatic vitals, adverse events assessment, physical exam) | 2 days
  Evaluation of orthostatic vitals signs, ECGs, and adverse event monitoring (Screening, Day -1, Day 1, Day 2), clinical lab testing and physical exam (Screening and Day 2)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Benesh, Study Director — Abbott

REFERENCES:
- [Result] Nyholm D, Odin P, Johansson A, Chatamra K, Locke C, Dutta S, Othman AA. Pharmacokinetics of levodopa, carbidopa, and 3-O-methyldopa following 16-hour jejunal infusion of levodopa-carbidopa intestinal gel in advanced Parkinson's disease patients. AAPS J. 2013 Apr;15(2):316-23. doi: 10.1208/s12248-012-9439-1. Epub 2012 Dec 11. PMID 23229334